CLINICAL TRIAL: NCT01986634
Title: Efficacy of Spot Treatment of Perioral Rhytids Compared to Full Field Laser Resurfacing
Brief Title: Laser Spot Treatment of Perioral Rhytids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 01-13-12
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Facial Aging
Keywords: Laser Resurfacing; Rhytids; Perioral
MeSH Terms: interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laser Treatment (Other): Patients enrolled will have split face laser treatment. Patients will serve as their own control.
  Interventions: Procedure: Laser Treatment

INTERVENTIONS:
Procedure: Laser Treatment — Patient will have split face laser resurfacing as per standard of care. One side of the face will be treated with a standardized single depth laser peel. The other side of the perioral area will be treated with variant, deeper treatment to perioral rhytids.

SUMMARY:
Perioral rhytides present a difficult problem in facial rejuvenation. They cannot be addressed with rhytidectomy (face lift) and direct excision can leave visible unfavorable scars. Currently, fine static wrinkles are most effectively treated with facial resurfacing, usually with laser treatment. Often the peri-oral area is treated with additional spot treatments with an ablative laser to cause a more robust healing response and better aesthtic result. To date, no studies have specifically shown efficacy of additional spot treatment over full facial laser alone.

This study is designed as a split-face study, to compare the aesthetic results of full field laser resurfacing on one half of the face with that of spot treatment of perioral rhytides on the other half.

To clarify further to the IRB board, this is not an experimental treatment. Spot treatment is used by many surgeons/laser proceduralists for addressing specific areas of the face. This is an FDA indicated use of the laser for facial resurfacing. Due to the many genetic and enviromental factors that can effect the results the best design for the study to is have each patient serve as their own control with a split-face study.

DETAILED DESCRIPTION:
Cohort Study, with Split Face treatment

Methods:

Patients will be evaluated in the office for possible inclusion. Those who agree to partipate will receive preoperative photos.

On the day of the procedure patients will have a topical anesthestic applied for 30 minutes, then patients will recieve a 20um laser resurfacing of the entire face to remove dead skin and debris. After that, patients will have reapplication of a topical anesthetic for an additional 10 minutes. They will then undergo a 50 um peel to one side of the face and a patient tailored spot treatment of perioral wrinkles to the other side of the face. The depth of this may vary from 100 to 400um.

Patients will return to clinic at 1 week, 2 weeks, and 3 weeks post-procedure and fill out a short survey and have medical photography done. Patients will return at 3 and 6 month follow-up for additional photography and surveys. These visits will typically take 10 to 20 minutes.

Preoperative and post-operative photos will be analyzed by 2 independent plastic surgeons for post-operative changes and improvements.

ELIGIBILITY:
Inclusion Criteria:

Patient who are electively presenting to the plastic surgery department for evaluation and treatment of facial aging and elect/seek to have laser treatment will be asked to voluntarily participate in the study.

Fitzpatrick type 1-4 skin

Exclusion Criteria:

1 Patients undergoing additional invasive cosmetic procedure at the same time including rhytidectomy, fat injection

2 History of Photosensitvity

3 Use of photosenstive medications

4 History of keloid or hypertrophic scarring

5 Use of Isotretinoin in the previous year

6 Previous resurfacing procedure (laser or chemical peel) within the previous 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Improvement in perioral rhytids | 3-6 months
  at 3 and 6 month post-operative visits, photographs will be taken and analyzed for improvement in rhytids.

SECONDARY OUTCOMES:
Time to healing after laser resurfacing | 2-3 weeks
  Each side of the face will be assessed for time to healing.

CONTACTS AND LOCATIONS:
Overall Officials: David J Rowe, MD, Principal Investigator — University Hospitals
Locations (1):
- Univeristy Hospitals Cedar Brainard Office, Lyndhurst, Ohio, United States